CLINICAL TRIAL: NCT02750865
Title: Conversational Agents to Improve Quality of Life in Palliative Care
Acronym: ECA-PAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Collaborators: Northeastern University (Other); Boston University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H-34877; 1R01NR016131 (NIH)
Record Dates: First submitted 2016-03-30; First posted 2016-04-26 (Estimated); Last update posted 2023-07-13 (Actual); Status verified 2023-07

CONDITIONS: Palliative Care
Keywords: biomedical technology; palliative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Usual Care (No Intervention): In this arm the subject receives usual care and just completes the baseline interview, monthly telephone surveys about their quality of life, and the exit interview at 6 months after enrollment.
- Embodied Conversational Agent (ECA) (Experimental): In this arm the subject is trained how to use a tablet device which they take home for the duration of the study. These subjects complete the baseline interview, monthly telephone surveys about their quality of life, and the exit interview at 6 months after enrollment.
  Interventions: Behavioral: Embodied Conversational Agent (ECA)

INTERVENTIONS:
Behavioral: Embodied Conversational Agent (ECA) — The ECA is a computer generated character who will interact with the subject on a daily basis via a touch-screen tablet. The system is designed to provide the following functions: (1) medication counseling; (2) physical activity promotion; (3) symptom management and continual screening for adverse events; and (4) alleviation of stress and anxiety. The investigators will augment the system to include: (5) spiritual needs assessment; and (6) advanced care planning.
  Arms: Embodied Conversational Agent (ECA)

SUMMARY:
In this study the investigators will advance research on the development of easy to use technologies to empower patients. This is a scalable approach that has a significant potential to reduce suffering for palliative care patients and their caregivers. The investigators will adapt existing tested empathic conversational agents (ECA) for home-based cancer care management and inpatient bedside counseling to provide the following functions:

1. medication counseling;
2. physical activity promotion;
3. symptom management and continual screening for adverse events; and
4. alleviation of stress and anxiety
5. spiritual needs assessment; and
6. advanced care planning.

Data from the system will be monitored by a health professional, who communicates with members of the patient's care team. In this project, this activity will include facilitating referral for palliative care services.

The investigators will conduct pilot studies both at Boston Medical Center and at Northeastern University that will test system usability (Northeastern University and BMC) as well as interview burden (BMC only).

The investigators will conduct a Randomized Control Trial (RCT) to evaluate the agent technology, comparing usual care (UC) versus usual care plus the agent (UC+ECA) for patients 21 or older, with a life expectancy of < 1 year, from outpatient clinics at Boston Medical Center (BMC). Each subject will be enrolled along with a caregiver surrogate subject. In addition to baseline data collection, there will be monthly phone surveys for six months; intervention subjects will use the system for a six-month period of time. In addition, the investigators will conduct a randomized trial within the intervention group to compare subjects getting functions 1-4 (above) versus subjects getting the augmented intervention with all six functions. The intervention will include a nurse management interface to monitor clinical alerts generated by the system to stimulate interventions by the clinical staff.

DETAILED DESCRIPTION:
Pilot Study The pilot study will determine usability of the ECA tablet system. Healthy volunteers will be recruited at Northeastern University, where the system is being developed. Subjects will spend approximately 60 minutes with the tablet system and provide usability feedback. Twelve healthy patient volunteers will be recruited to review the system as well as provide feedback on the relative interview burden (was the interview too long, too invasive, etc). No identifiable data will be collected from pilot study subjects.

Main Study The study will consist of adults with advanced illness (health care provider endorses the existence of a potentially life-limiting condition and endorses that "it would not be a surprise if the patient died within 12 months") who will be randomized to intervention or usual care control groups. Each person with an advanced illness will be enrolled along with a caregiver (i.e., family, friend) who will serve as a surrogate subject. The caregiver will be consented at baseline and interviewed at that point and at the final, 6-month study visit. In addition, if, at any point during their enrollment in the study, the patient-subject becomes unable, or decisionally impaired, to answer interview questions, the caregiver will be asked to answer on behalf of the subject.

The patient can be found to be decisionally impaired in any of 3 ways:

1. the patient declares themselves to be unable to answer questions appropriately
2. the patient is unable to pass a brief cognitive assessment that will be administered at the beginning of each telephone follow-up (per the Brief Screen for Cognitive Impairment)
3. the patient is physically unable to answer questions on the phone (due to, for example, serious health decline or death)

Baseline data will be collected after enrollment and before randomization. Baseline data includes:

1. sociodemographic data
2. Quality of life as measured by the European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire-Palliative Care
3. Patient Reported Outcomes Measurement Information System (PROMIS) Mental Health
4. Patient Reported Outcomes Measurement Information System (PROMIS) Social Health
5. Patient Activation Measure (PAM)
6. Patient Medication Adherence Questionnaire (PMAQ)
7. Spiritual Needs Assessment for Patients (SNAP)
8. Community Healthy Activity Model Program for Seniors (CHAMPS)
9. a survey of Advance Care Planning (ACP) communication and preferences
10. BSCI (This cognitive assessment is non-exclusionary, but, if the patient scores "0" on the word recall, the designated caregiver/surrogate will be asked to act as the research proxy and answer questions for the patient-subject.)

The investigators will also interview the surrogate subject at baseline regarding their level of caregiver stress with:

1. the CarerQol-7D
2. the caregiver's level of happiness (CarerQol-VAS)
3. self-rated burden (SRB) of care giving After the initial visit, study staff will administer 5 monthly phone surveys (months 1, 2, 3, 4, and 5), where the EORTC QLQ-C15-PAL will be collected. At the beginning of each data collection point study staff will administer the Brief Survey of Cognitive Impairment (BSCI) to determine if the patient is cognitively able to answer questions, and also inquire about unplanned health care utilization (i.e., urgent care, emergency room, hospital observation visits, and hospital admissions).

At the final, 6-month visit, the patient-subject will be interviewed in person, with the surrogate, and the full list of instruments will be administered. In addition, study staff will prepare a summary data report for the patient's clinical team. The report will include obtaining information from the Palliative Care service. The research staff will ask the subject which clinicians of theirs they would like to have receive this information.

Subjects randomized to the intervention will be given a mini-tablet computer configured for the purposes of this study. A research assistant will set up the tablet, enroll subjects into the study database, and train these subjects in the use of the system. Subjects who do not have existing WiFi at home will be provided with a cellular-based router. In such cases, study staff will arrange the WiFi service plan, install the router in the home, and confirm connectivity.

The investigators estimate that in many instances, when a clinician endorses that they would not be surprised if their patient died within 12 months, that this would be the first time they solidified a prognostic outlook in their minds for that patient. Stimulating clinicians to consider their patient's life-expectancy is itself a form of intervention, as this may instigate communication about prognosis with the patient, a re-evaluation of the treatment course, assessment of goals of care, and an improved level of attention to symptoms. The investigators will conduct informational sessions about the study and provide material about palliative care services in each outpatient clinical environment from which subjects will be enrolled. Information will be provided on how clinicians can contact the Palliative Care service to obtain consultation. Clinicians will be encouraged to call for assistance on palliative care needs for intervention subjects, usual care subjects, and non-subjects.

The same measures collected at baseline will also be collected at the final 6-month interview. At the end of study participation the investigators will also prepare a summary data report for the patient's clinical team. The report will include information on obtaining consultation from the Palliative Care service. The research nurse will ask the subject which clinicians of theirs they would like to have receive this information.

ELIGIBILITY:
Inclusion Criteria:

1. 21 years of age or older
2. English speaking
3. Able to independently consent to be in the study
4. Has adequate corrected vision to be able to use the ECA system (based on a 1-minute ECA functional screener)
5. Has adequate hearing to be able to use the ECA system (headphones will be available)
6. Has a health care provider who endorses the existence of a potentially life-limiting condition and endorses that it would not be a surprise if the patient died within 12 months (PATIENT-SUBJECTS only)

Exclusion Criteria:

1. Enrolled in hospice
2. Already being followed by the Palliative Care team
3. Suicidal or homicidal
4. In police custody
5. Do not live in the Boston area
6. Plan on leaving the Boston area for more than 4 weeks in the next 6 months
7. Not able to use the ECA tablet computer

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 367 (Actual)
Dates: Start 2017-08-02 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Quality of Life of palliative cancer care participants | assessed monthly up to 6 months
  QOL will be assessed using QLQ-C15-PAL, a 15-scale-item instrument designed to assess the quality of life of participants.

SECONDARY OUTCOMES:
Palliative Care services utilization | assessed monthly up to 6 months
  Rate of receiving palliative care services as evidenced by presence of at least one Palliative Care clinical note in the EMR.
Hospital utilization | assessed at 6 months
  Data on healthcare utilization will be obtained through EMR review and monthly phone survey of all subjects for six months, or until patient death. The investigators will obtain data on the number of urgent care, emergency room, hospital observation visits, and hospital admissions.
Cost | assessed at 6 months
  Costs will be obtained from the actual observed costs from the annual Medical Expenditure Panel Surveys (MEPS) conducted the Agency for Healthcare Research and Quality (AHRQ), specific to each service type (ED, inpatient stay and outpatient visit) and reason for visit (principal diagnosis). We will also adjust for inflation in costs over time. The primary utilization measure will be the total costs for all ED visits, inpatient stays, and outpatient physician visits. As secondary measures the investigators will examine the cost of different services. As a simple budget impact assessment the investigators will also evaluate the cost of the intervention, specifically, the provision of additional nurse management services.
Mental health | assessed at enrollment and at 6 months
  Mental and Social health will be assessed using the PROMIS Mental Health (including subscales on: depression, anxiety, anger, cognitive function, alcohol use, consequences, and expectancies, psychosocial illness impact, self-efficacy, and smoking,) and PROMIS Social Health (including subscales on: ability to participate in social roles and activities, satisfaction with social roles and activities, social support, social isolation, and companionship) instruments. The NIH PROMIS measures have been subjected to extensive reliability and validity testing.
Patient activation | assessed at enrollment and at 6 months
  Patient Activation will be measured using the Patient Activation Measure (PAM).
Medication adherence | assessed at enrollment and at 6 months
  Medication Adherence will be assessed using the Patient Medication Adherence Questionnaire (PMAQ).
Symptoms | assessed at enrollment and at 6 months
  Symptoms will be assessed using the Edmonton Symptom Assessment Scale-revised (ESAS-r).
Spiritual Needs | assessed at enrollment and at 6 months
  Spiritual Needs will be assessed using the Spiritual Needs Assessment for Patients instrument (SNAP). SNAP includes 23 items in three domains: psychosocial (n=5), spiritual (n=13), and religious (n=5).
Medical Orders for Life-Sustaining Treatment (MOLST) completion rate | assessed at enrollment and at 6 months
  MOLST form completion rate as identified in the Electronic Medical Record
Advance Care Planning and preferences | assessed at enrollment and at 6 months
  ACP communication and preferences will be assessed using a survey that the investigators have used in prior work.
Physical activity | assessed at enrollment and at 6 months
  Physical activity will be assessed using the walking items from the validated CHAMPS questionnaire for older adults. The CHAMPS assesses usual weekly amounts of walking over the previous 4 weeks in minutes per week, and these items have been significantly associated with pedometer steps and were sensitive to change with a prior ECA-based walking promotion intervention for older adults.
Use of the ECA-PAL system by subjects in the intervention group | assessed at 6 months
  Use of the ECA-PAL system will be determined from log files stored in the database, describing the details of all sessions with the patients, including all discussion topics and questions asked.
Satisfaction with the ECA-PAL system | assessed at 6 months
  Satisfaction with the ECA-PAL system will be assessed using attitudinal measures that have been used in the investigators' prior work. These include the 19-item computer program acceptability scale, and the 12-item bonding subscale of the Working Alliance Inventory (WAI).
Social health | assessed at enrollment and at 6 months
  Social health will be assessed using the PROMIS Social Health (including subscales on: ability to participate in social roles and activities, satisfaction with social roles and activities, social support, social isolation, and companionship) instruments.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Dedier, MD, Principal Investigator — Boston Medical Center; Michael Paasche-Orlow, MD, MPH, Principal Investigator — Tufts Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT02750865/ICF_000.pdf